CLINICAL TRIAL: NCT04561440
Title: Copy Number Variation in Prenatal Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: YiYang Zhu (Other)
Responsible Party: Sponsor-Investigator, YiYang Zhu, vice dean of prenatal dignosis, Taizhou Hospital
Organization: Taizhou Hospital (Other)
Other Study IDs: 19EZZDC7
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Copy Number Variation; Genome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- molecular karyotyping
  Interventions: Diagnostic Test: molecular karyotyping
- cytogenic karyotyping
  Interventions: Diagnostic Test: molecular karyotyping

INTERVENTIONS:
Diagnostic Test: molecular karyotyping — performed by NGS or CMA chip

SUMMARY:
An observed study is aim to map the CNVs distribution in human genome of Chinese prenatal population.

Setting: Prenatal diagnosis center of Taizhou City, Zhejiang Province Patient: total cases of pregnant women needed prenatal genetic diagnosing Methods: karyotype was performed with combined of molecular and cytogenic protocol. Subgroup: molecular karyotyping performed by genomic Chip (CMA) or NGS, the latter including cnv-seq and NIPT.

Main outcome: comparison of CNVs distributions in subgroups. Second outcome: comparison of CNVs distributions in demographic dates.

ELIGIBILITY:
Inclusion Criteria:

* total population need invasival prenatal diagnosis

Exclusion Criteria:

* multipara

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: total population need invasival prenatal diagnosis, which including total pregnant women whose aged over than 35 in Taizhou City of East China.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
comparison of CNVs distributions in subgroups | 2016-2020
  subgroups including CNV-seq (by NGS) and CMA chip

SECONDARY OUTCOMES:
comparison of CNVs distributions in demographic dates. | 2016-2020
  demographic dates including indication of prenatal diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Taizhou Hospital of Zhejiang province, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided